CLINICAL TRIAL: NCT03417167
Title: "Interest of Synovial Biopsy in the Etiological Assessment of Arthritis of Undetermined Origin: Multicenter Prospective Series"
Brief Title: Indications and Interest of US-guided Synovial Biopsies Performed in Clinical Practice
Acronym: BIOPSYN
Status: Completed | Type: Observational
Sponsor: Nantes University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: RC17_0440
Record Dates: First submitted 2018-01-15; First posted 2018-01-31 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2018-01

CONDITIONS: Arthritis
Keywords: synovial biopsy; US guided synovial biopsy
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: US-guided synovial biopsy — Needle Synovial biopsy performed using a Tru-cut® device.

SUMMARY:
Synovial biopsies are now routinely performed both in research and in clinical practice. The developments of ultrasound (US) and of US-guided needle biopsies devices have facilitated their use and tolerance by the patients. However, their interest in clinical practice in the context of an undifferentiated arthritis remains debated.

DETAILED DESCRIPTION:
In this study, the investigators will collect all the synovial biopsies performed in clinical practice in 18 Rheumatology Unit throughout France. All the participants received a standardized training on US-guided synovial biopsies. For each biopsy, the indications, clinical presentation, procedure (length, tolerance), biopsy results (Pathology, bacteriology, etc ...) will be collected in a Clinical Research Form. The investigator will determine the number of cases where the synovial biopsy allows drawing a definite diagnosis.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing an US-guided synovial biopsy in clinical practice in the context of an arthritis of unknown origin

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Age under 18 year old, pregnancy, breastfeeding
Sampling Method: Non-Probability Sample
Enrollment: 201 (Actual)
Dates: Start 2018-02-14 (Actual); Primary Completion 2020-09-11 (Actual); Study Completion 2020-09-11 (Actual)

PRIMARY OUTCOMES:
number of cases where the synovial biopsy allows drawing a definite diagnosis | 10 days
  Final diagnosis will be classified in 5 groups: infectious, crystal induced arthritis, tumoral, inflammatory rheumatisms, others (amyloidosis etc …)

SECONDARY OUTCOMES:
Indications, tolerance, complications, number and type of analysis for each sample, results of pathology, bacteriology, mycobacteriology | 1 month
  For each biopsy, the indications, clinical presentation, procedure (length, tolerance), biopsy results (Pathology, bacteriology, etc ...) will be collected in a Clinical Research Form.

CONTACTS AND LOCATIONS:
Overall Officials: Benoit Le Goff, Principal Investigator — Nantes University Hospital
Locations (17):
- France (17):
  - AP-HP, Paris, Lariboisière
  - AP-HP, Paris, Saint-Antoine
  - AP-HP, Paris, Salpétrière
  - Chu d'Angers, Angers
  - CHU de Bordeaux, Bordeaux
  - Chu Brest, Brest
  - CHU CAEN, Caen
  - Chu de Dijon, Dijon
  - CHD La Roche-sur-Yon, La Roche-sur-Yon
  - AP-HM, Marseille
  - Chu de Montpellier, Montpellier
  - CHU de Nancy, Nancy
  - CHU de Nice, Nice
  - CHU de Poitiers, Poitiers
  - Chu de Rennes, Rennes
  - Chu de Strasbourg, Strasbourg
  - Chu de Toulouse, Toulouse